CLINICAL TRIAL: NCT00344669
Title: Increased Weight Gain in Preschool Children Due to Mass Albendazole Treatment Given During "Child Health Days" in Uganda
Brief Title: Effect of Mass Deworming on Child Growth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makerere University (Other)
Collaborators: Ministry of Health, Uganda (Other Government); World Bank (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P05267
Record Dates: First submitted 2006-06-14; First posted 2006-06-27 (Estimated); Last update posted 2006-10-17 (Estimated); Status verified 2006-06

CONDITIONS: Low Weight for Age in Preschool Children
Keywords: underweight; preschool; mass deworming
MeSH Terms: conditions — Thinness | interventions — Albendazole

INTERVENTIONS:
Drug: Albendazole 400 mg, given 6 monthly

SUMMARY:
The purpose of the study was to determine whether periodical mass deworming improves growth in children below six years of age.

DETAILED DESCRIPTION:
Many children in developing countries get slowed growth because of heavy loads of intestinal helminths. Quite often treatment is not sought because there may not be any obvious symptoms. Slowed growth may manifest as low weight for age or low height for age.

The objective of the study was to estimate the effectiveness of the delivery of an anthelmintic drug through a community child health program on the weight gain of preschool aged children.

Design: This was a cluster randomized controlled trial in 48 parishes in Eastern Uganda. All 48 parishes were participating in a new program for child health; 24 were randomly assigned to offer to children an additional service of anthelmintic treatment. The intervention was 400 mg of albendazole added to the standard services at child days over a 3 years period. All children were offered the drug and the main outcome measure was weight gain.

Results: A total of 27,995 children were recruited into the 2 arms of the study with 14,940 in the treatment arm and 13,055 in the control arm. The intervention arm got an increase in weight gain of about 10% (166 grams per child per year (CI: 16-316) above expected weight gain when treatment was taken twice a year and an increase of 5% when treatment was received approximately annually.

Conclusion: The inclusion of deworming in regularly scheduled health services appears practical and capable of increasing child growth.

ELIGIBILITY:
Inclusion Criteria:

* children 1-6 years

Exclusion Criteria:

-

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10000
Dates: Start 2000-08; Study Completion 2003-11

PRIMARY OUTCOMES:
weight gain
weight for age

CONTACTS AND LOCATIONS:
Overall Officials: Joseph K Konde-Lule, MD DPH MSc, Principal Investigator — Makerere University; John F Mutumba, MBChB, MSc, Study Chair — Ministry of Health, Uganda
Locations (1):
- 48 parishes in Eastern Uganda, Kampala, Uganda